CLINICAL TRIAL: NCT05357001
Title: Effects of Connective Tissue Manipulation Versus Stretching Exercises on Pain and Symptoms Severity in Females With Primary Dysmenorrhea
Brief Title: Effects of Connective Tissue Manipulation Versus Stretching Exercises in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0501
Record Dates: First submitted 2022-04-15; First posted 2022-05-02 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary dysmenorrhea; Connective tissue manipulation; Stretching
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue manipulation (Experimental): technique to remove muscle spasticity
  Interventions: Other: Connective tissue manipulation
- stretching exercise (Experimental): exercises to remove muscle spasticity
  Interventions: Other: stretching exercises

INTERVENTIONS:
Other: Connective tissue manipulation — to remove muscle spasticity
  Arms: Connective tissue manipulation
Other: stretching exercises — to remove muscle spasticity
  Arms: stretching exercise

SUMMARY:
The study will be a randomized clinical trial in which the effect of connective tissue manipulation will be compared with the effect of stretching exercises on pain and severity of symptoms in primary dysmenorrhea. Inclusion criteria will include nulliparous females in the age range of 18-25 years old. Exclusion criteria will be women with irregular menses (<21 and >35 days), systemic and gynecological diseases (gastrointestinal, autoimmune, psychiatric diseases, endometriosis, pelvic inflammatory diseases), pregnant women, previous pelvic surgery, traumatic injury. The participants will be allocated to two groups, group A and B. Group A will receive connective tissue manipulation on sacral, lumbar, lower thoracic and anterior pelvic regions with the patient in sitting and supine positions. Group B will receive active stretching exercise regime including forward, backward ad side trunk bending, heel raise, half squatting, knee to chest, hamstring stretching, calf stretching and abdominal contractions.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial in which the effect of connective tissue manipulation will be compared with the effect of stretching exercises on pain and severity of symptoms in primary dysmenorrhea. Inclusion criteria will include nulliparous females in the age range of 18-25 years old. Exclusion criteria will be women with irregular menses (<21 and >35 days), systemic and gynecological diseases (gastrointestinal, autoimmune, psychiatric diseases, endometriosis, pelvic inflammatory diseases), pregnant women, previous pelvic surgery, traumatic injury. The participants will be allocated to two groups, group A and B. Group A will receive connective tissue manipulation on sacral, lumbar, lower thoracic and anterior pelvic regions with the patient in sitting and supine positions. Group B will receive active stretching exercise regime including forward, backward ad side trunk bending, heel raise, half squatting, knee to chest, hamstring stretching, calf stretching and abdominal contractions.

All the participants will be informed about the manner of research and will be asked to sign the consent form after they are willing to participate in the study. WaLIDD score and dysmenorrhea severity scoring will be used to determine and assess the dysmenorrhea pain and severity. Treatment sessions will be conducted for 8 weeks, 3 times in a week and each session will be carried out for 20 minutes. At the end of two months, subjects will be assessed for their two menstrual cycles. SPSS 21 will be used for data analysis. After checking normality of data appropriate tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women • Age range of 18 to 25 years

Exclusion Criteria:

* Women with irregular menses (<21 days and >35 days)
* Systemic and gynecological diseases
* Pregnant women
* Women taking contraceptive pills
* Traumatic injuries
* Previous pelvic surgery

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female only
Enrollment: 22 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
WaLIDD | 6 months
  WaLIDD (Working ability, location, intensity, days of pain, dysmenorrhea) score and dysmenorrhea severity score.
  It was designed, which integrated features of dysmenorrhea such as:
  1. number of anatomical pain locations (no part of the body, lower abdomen, lumbar region, lower limbs, inguinal region),
  2. Wong-Baker pain range (does not hurt, hurts a little, hurts a little more, hurts even more, hurts a lot, hurts a lot more),
  3. number of days of pain during menstruation (0, 1-2, 3-4, ≥5), and
  4. frequency of disabling pain to perform their activities (never, almost never, almost always, always).
  Each tool's variable provided a specific score between 0 and 3, and the final score ranged from 0 to 12 points
  Score: 0 without dysmenorrhea, 1-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 severe dysmenorrhea. Wong-Baker scale was reclassified to adjust a four-level scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabiya Noor, PhD, Study Chair — Riphah International University
Locations (1):
- Jinah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osuga Y, Hayashi K, Kanda S. Long-term use of dienogest for the treatment of primary and secondary dysmenorrhea. J Obstet Gynaecol Res. 2020 Apr;46(4):606-617. doi: 10.1111/jog.14209. Epub 2020 Feb 12. PMID 32050307
- [Background] Osayande AS, Mehulic S. Diagnosis and initial management of dysmenorrhea. Am Fam Physician. 2014 Mar 1;89(5):341-6. PMID 24695505
- [Background] Habibi N, Huang MS, Gan WY, Zulida R, Safavi SM. Prevalence of Primary Dysmenorrhea and Factors Associated with Its Intensity Among Undergraduate Students: A Cross-Sectional Study. Pain Manag Nurs. 2015 Dec;16(6):855-61. doi: 10.1016/j.pmn.2015.07.001. Epub 2015 Aug 29. PMID 26328887